CLINICAL TRIAL: NCT05268744
Title: Micronutrient Supplementation in Children With Autism Spectrum Disorder (ASD): A Clinical Trial Examining Mechanism of Action
Brief Title: Micronutrient Supplementation in Children With ASD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-35971
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Micronutrients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Micronutrient (Experimental): In this open-label trial, all subjects will receive the daily dose of micronutrient, in the form of one lightning stick per day, which contains 2.9 grams of micronutrients per stick. It will be delivered in a powder form taken sublingually.
  Interventions: Drug: Micronutrient

INTERVENTIONS:
Drug: Micronutrient — Subject will take micronutrient supplement daily for 8 weeks

SUMMARY:
An open-label examination of changes in metabolites with use of micronutrients in children with autism spectrum disorder (ASD). Investigators will also measure behavioral measures monthly at school with teachers and parents report.

DETAILED DESCRIPTION:
Children enrolled in Oak Hill School will enroll in this study and take micronutrient supplement once a day for 8 weeks period. Behavioral measures and metabolites taken from Dried Blood Spots (DBS) will be collected pre and post treatment. Behavioral measures will be taken again at 12 weeks, after 4 weeks of not dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, enrolled at Oak Hill School (OHS), age 6-22 and with a diagnosis of ASD.
2. ASD diagnosis will be established by standard criteria (DSM-IV criteria and expert clinician review of medical records and child observation).
3. Written informed consent obtained from the subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. Taking multivitamins currently and unwilling to stop during the study period

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hendren, DO, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants received the daily dose of micronutrient, in the form of one lightning stick per day, which contains 2.9 grams of micronutrients per stick. It was delivered in a powder form and taken sublingually.
Period: Overall Study
Arm/Group | All Participants
Started | 16
Completed | 11
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Autism Behavior Inventory - Short (ABI-S) [Mean (Standard Deviation); unit: units on a scale]
  ABI-S (Parent) | 25.3 (3.5)
  ABI-S (Teacher) | 21.6 (10.7)
Social Responsiveness Scale (SRS) [Mean (Standard Deviation); unit: units on a scale]
  SRS (Parent) | 94.4 (23.8)
  SRS (Teacher) | 69 (24.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Autism Behavior Inventory, Short Form (ABI-S)
Description: The ABI-S is an observer-reported outcome scale designed specifically to measure change and severity of Autism Spectrum Disorder (ASD) symptoms. ABI-S will be measured by both parents and teachers. There are 24 questions. The scoring of ABI-S questions can range from 0-3 (with possible reverse scoring) based on scoring instructions for data analysis. The total range of score is between 0 and 72. Lower score indicates better performance.
Time Frame: Baseline to Week 8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 11
score on a scale
  ABI-S (Parent) | -2.9 [-7.1 to 1.4]
  ABI-S (Teacher) | -0.8 [-4.4 to 2.8]
Statistical Analysis 1: Comparison: All Participants; Null hypothesis was no improvement in mean ABI-S and SRS scores at the end of the study, compared to baseline; Test type: Superiority — Since all outcomes were normally distributed, one-sided paired t-test was used to compare mean pre- and post-treatment scores to see whether post-treatment scores of ABI-S and SRS had improved compared to pre-treatment scores; p < 0.05, t-test, 1 sided

2. Primary Outcome: Change in the Social Responsiveness Scale (SRS)
Description: SRS measures social ability in children and young adults. SRS will be measured by both parents and teachers. There are 65 questions. The scoring of SRS questions can range from 0-3 (with possible reverse scoring) based on scoring instructions for data analysis. The total possible score range for the SRS is 0 - 195. Lower score indicates better performance.
Time Frame: Baseline to Week 8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 11
score on a scale
  SRS (Parent) | -8.1 [-18.4 to 2.2]
  SRS (Teacher) | 0.8 [-9.8 to 11.4]

ADVERSE EVENTS:
Time Frame: 8 Weeks
Groups:
- All Study Participants: All Participants with ASD enrolled in the 8-week open-label study of micronutrient supplements.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
The limited sample size (N=11) has indeed constrained the statistical power of the analysis.

The absence of a control group prevents direct comparisons between treated participants and untreated individuals, limiting our ability to isolate the effects of the micronutrient supplement from other confounding factors.

We do not have information regarding the types of diets the participants were on which could have influenced their response to the micronutrient supplementation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT05268744/Prot_SAP_000.pdf